CLINICAL TRIAL: NCT05014464
Title: Molecular Characterization and Clinical Outcomes of ALK Tyrosine Kinase Inhibitors in ALK-rearranged Advanced Squamous Cell Carcinoma
Brief Title: ALK Tyrosine Kinase Inhibitors in ALK-rearranged Advanced Squamous Cell Carcinoma
Acronym: ATPase
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210119
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ALK rearrangement; Squamous cell lung cancer; ALK-TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; alectinib; brigatinib; lorlatinib; Pemetrexed; Immune Checkpoint Inhibitors; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A, first line ALK-TKIs (Experimental): All the patients were treated with first line ALK-TKis including Crizotinib, Alectinib, Brigatinib and Lorlatinib etc. Approximately 30 patients.
  Interventions: Drug: Crizotinib
- Cohort B, second line ALK-TKIs (Experimental): All the patients were treated with second line ALK-TKis including Crizotinib, Alectinib, Brigatinib and Lorlatinib etc. Approximately 30 patients.
  Interventions: Drug: Crizotinib
- Cohort C, post second line ALK-TKIs (Experimental): All the patients were treated with post second ALK-TKis including Crizotinib, Alectinib, Brigatinib and Lorlatinib etc. Approximately 30 patients.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib 250mg po bid Aectinib 600mg po bid Lorlatinib 100mg po qd Brigatinib, 90mg po qd for one week and than 180mg po qd forever Pemetrexed 500mg/m2
  Other Names: Alectinib; Brigatinib; Lorlatinib; Pemetrexed; immune checkpoint inhibitors; Carboplatin; Paclitaxel

SUMMARY:
This study was to explore the efficacy of ALK-TKI in lung squamous cell carcinoma. Approximately 5% of lung adenocarcinomas have oncogenic fusions of EML-4 and ALK a mutation associated with tumorigenesis and migration.

DETAILED DESCRIPTION:
This research focuses on exploring epidemiology, distributions and the efficacy and prognosis of ALK-TKI in lung squamous cell carcinoma.Approximately 5% of lung adenocarcinomas have oncogenic fusions of EML-4 and ALK a mutation associated with tumorigenesis and migration. Several studies have shown that in patients with ALK-rearranged non-small cells, the use of ALK inhibitors can achieve better efficacy and significantly prolong overall survival. However few of them performed Fish or NGS tests. Our data demonstrates that lung squamous cell carcinoma with ALK rearrangement responds well to ALK-TKI, and correspondingly has a significant improvement in survival time and prognosis, providing a basis for the treatment of ALK-positive patients with lung squamous cell carcinoma. At the same time, we believe that genetic testing is also required for lung squamous cell carcinoma to achieve more accurate medication.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histopathology or cytology confirmed and recorded local progression or metastatic Advanced Squamous Cell Carcinoma without systemic treatment.
4. ALK fusion positive evaluated by IHC (ventana), NGS or FISH.
5. ECOG 0 - 1.
6. Predicted survival ≥ 12 weeks.
7. Adequate bone marrow hematopoiesis and organ function
8. Presence of measurable lesions according to RECIST 1.1.
9. Subjects with stable brain metastases may be included in the study.

Exclusion Criteria:

1. Prior systemic therapy for locally advanced or metastatic disease.
2. Subjects who have received any of the following treatments must be excluded:

   * Treatment with molecules such as EGFR, VEGFR antibodies within 4 weeks prior to the first dose of study drug.
   * Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
   * Ongoing (or inability to discontinue) possibly potent CYP1A2, CYP3A inhibitor (1 week), or inducer (2 weeks) drug therapy or herbal supplements within 1-2 weeks prior to the first dose.
3. Presence of spinal cord compression or meningeal metastasis.
4. History of other malignant tumors within 2 years.
5. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
8. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
9. Heart-related diseases or abnormalities
10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
12. Live vaccine was given 2 weeks before the first medication.
13. Women who are breastfeeding or pregnant.
14. Hypersensitivity to the test drug and the ingredients.
15. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-08-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated by different treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause

SECONDARY OUTCOMES:
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 month.
  To assess overall survival, define as first dose to the death of the subject due to any cause
Objective Response Rate (ORR) | Time from first dose to last dose, or up to 24 month.
  To assess ICI and TKIs overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China